CLINICAL TRIAL: NCT05919459
Title: Effectiveness of Acceptance and Commitment Therapy Versus Active Controls in Improving Psychological Functions of Parents and Children With Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20221121001
Record Dates: First submitted 2023-05-30; First posted 2023-06-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis (AIS); Acceptance and commitment therapy (ACT); parental psychological flexibility; psychological function; Randomized Controlled Trial (RCT)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parents with ACT intervention (Experimental): 5-week online synchronous ACT intervention plus asynchronous online AIS education
  Interventions: Behavioral: 5-week online synchronous ACT intervention; Behavioral: asynchronous online AIS education
- Parents without ACT intervention (Other): 5-week interactive online AIS education
  Interventions: Behavioral: asynchronous online AIS education

INTERVENTIONS:
Behavioral: 5-week online synchronous ACT intervention — Parents will meet a trained ACT counsellor to undergo five weekly sessions of ACT group training via Zoom. Specifically, each 120-minute synchronous videoconferencing session will involve the ACT counsellor and 6-8 parents.
  Arms: Parents with ACT intervention
Behavioral: asynchronous online AIS education — A healthcare educator with a background in nursing, physiotherapy, or occupational therapy will meet with parents in five weekly 120-minute interactive AIS-related education videoconferencing via Zoom. Specifically, each 120-minute synchronous videoconferencing session will involve the ACT counsellor and 6-8 parents.

SUMMARY:
Systematic reviews revealed that Acceptance and Commitment Therapy (ACT) for parents had medium-to-large effect sizes in improving parental depression/anxiety (d > 0.50), dysfunctional parenting styles (ds = 0.61-0.77), and small-to-large effect sizes in improving children's behavioral and emotional problems (ds = 0.25-0.84) in children/teenagers with various chronic diseases. A recent randomized controlled trial (RCT) showed that a web-based ACT program involving a coach providing semi-structured written feedback was significantly better than waitlist controls in improving the self-reported depression, anxiety, burnout, and psychological flexibility skills in parents of children/teenagers with chronic conditions (e.g., type 1 diabetes) up to 4 months post-treatment. The investigator's RCT also found that 4 weekly sessions of group-based ACT plus asthma education was significantly better than asthma education alone in improving parental psychological function (i.e., stress, anxiety, guilt, worries, sorrow, anger, and psychological flexibility), and participants' children's asthma symptoms at 6-month follow-up. The investigator's path analysis showed that ACT improved parental psychological flexibility, which mediated the decrease in parental distress and childhood asthma symptoms. These findings support that ACT for parents not only improves parental psychological flexibility and psychological controls, but also enhances social/emotional functioning of children/teenagers with different problems (e.g., chronic pain). Given the busy schedule of schoolchildren in Hong Kong and the promising results of ACT in improving the psychosocial well-being of both parents and teenagers, providing ACT to parents of teenagers with adolescent idiopathic scoliosis (AIS) may be a "killing two birds with one stone" solution to benefit both parents and teenagers. The current study will investigate this possibility.

DETAILED DESCRIPTION:
This is a single-blinded 2-arm RCT. A total of 168 parent-child dyads will be recruited consecutively from the scoliosis clinic in the Duchess of Kent Children's Hospital (DKCH). Eligible parents with the children will complete the baseline questionnaires and be randomized to either ACT or control group. Parents in the ACT group will be invited to join a 30-minute small private online course (SPOC) related to AIS. Parents in the ACT group will receive five weekly online ACT group-training sessions through Zoom. The controls will receive five weekly interactive online lectures/meetings through Zoom that will cover detailed topics related to AIS information and management. A research assistant, blinded to the group allocation, will use phone calls and emails to remind all participating parents and children to complete a set of online questionnaires identical to the baseline questionnaires at 5-, 12-, and 24-week follow-ups.

ELIGIBILITY:
Inclusion Criteria of 168 parent-child dyads:

1. the parent/guardian (henceforth "parents") aged between 25 and 60 years who is mainly responsible for taking care of a child with AIS (including the scoliosis clinic follow-ups)
2. the parent/guardian demonstrate at least mild anxiety (General Anxiety Disorder Scale scores > 5) or mild depressive symptoms (Patient Health Questionnaire scores > 5).
3. the parent/guardian live with the index child aged between 10 and 17 years.
4. the children have an orthopedist's diagnosis of AIS (Cobb angles of the major curve > 10º).
5. the children are managed conservatively or waiting for surgery scheduled more than six months later.
6. both parents and children should reside in Hong Kong for at least another six months.
7. both parents and children should be able to read/understand Chinese,
8. both parents and children can be reachable via phone/email, and can access the Internet on their own computers, tablets, or smartphones.

Exclusion Criteria:

1. parents and/or children with psychological disorders or behavioral problems (e.g., attention deficit hyperactivity disorder) that require regular psychological/psychiatric interventions;
2. children having undergone surgeries unrelated to AIS; or children with other types of scoliosis, or congenital diseases.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 336 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in self-report anxiety levels of the parent and child participants at 5-week follow-up | Baseline, 5-week follow-ups
  The 7-item Chinese version of the Generalized Anxiety Disorder scale (GAD-7) will be used to evaluate the self-report anxiety levels of the parent and child participants. It evaluates the severity of seven core-anxiety items in the previous two weeks.
Change from Baseline in severity of depression symptoms in the parent and child participants at 5-week follow-up | Baseline, 5-week follow-ups
  The 9-item Chinese version of the Patient Health Questionnaire (PHQ-9) will be used to measure the severity of depression symptoms in the parent and child participants. The items evaluate whether the symptoms have affected an individual in the previous 2 weeks.

SECONDARY OUTCOMES:
Change in stress level of the parent-child dyads | Baseline, 5-, 12-, and 24-week follow-ups
  The Chinese version of the Perceived Stress Scale-10 (PSS-10) will be used to assess the stress level of the parent-child dyads. The PSS-10 has good validity and reliability.
Change in parental psychological flexibility | Baseline, 5-, 12-, and 24-week follow-ups
  The 7-item Chinese version of the Acceptance and Action Questionnaire II (AAQ-II) will be used to measure parental psychological flexibility.
Change in family functioning for both parent and teen participants | Baseline, 5-, 12-, and 24-week follow-ups
  The 36-item Chinese version of the Self-report Family Inventory (C-SFI) will be administered to both parent and teen participants to evaluate the family functioning. C-SFI discerns dysfunctional families from competent ones. It has demonstrated high internal consistency and temporal stability in local families over 1 year.
Change in dysfunctional parenting styles in parents | Baseline, 5-, 12-, and 24-week follow-ups
  The 7-item Parenting Scale (PS-7) will be used to evaluate two dysfunctional parenting styles (over-reactivity [4 items] and laxness [3 items]) in parents. The factor score is the average score of the items in that factor. PS-7 has demonstrated good internal consistency and validity.
Change in parental caring burden level | Baseline, 5-, 12-, and 24-week follow-ups
  The Chinese version of 22-item Zarit Caregiver Burden Inventory (ZCBI) will be used to assess the parental caring burden level in health, mental state, social life, and finance. The questionnaire has demonstrated good internal consistency.
Change in teenager's health-related quality of life | Baseline, 5-, 12-, and 24-week follow-ups
  The Chinese version of the Scoliosis Research Society-22 (SRS-22r) questionnaire will be used to evaluate teenager's health-related quality of life (HRQOL). It comprises 22 questions in 5 domains: pain (5 items), self-image/appearance (5 items), mental health (5 items), function/activity (5 items), and satisfaction with management (2 items). Each item is graded on a 5-point scale ranging from 1 to 5. Higher scores indicate better HRQOL. The SRS-22r has demonstrated high reliability and validity in local adolescents.
Change from Baseline in self-report anxiety levels of the parent and child participants at 12-, and 24-week follow-ups | Baseline,12-, and 24-week follow-ups
  The 7-item Chinese version of the Generalized Anxiety Disorder scale (GAD-7) will be used to evaluate the self-report anxiety levels of the parent and child participants. It evaluates the severity of seven core-anxiety items in the previous two weeks.
Change from Baseline in severity of depression symptoms in the parent and child participants at 12-, and 24-week follow-ups | Baseline, 12-, and 24-week follow-ups
  The 9-item Chinese version of the Patient Health Questionnaire (PHQ-9) will be used to measure the severity of depression symptoms in the parent and child participants. The items evaluate whether the symptoms have affected an individual in the previous 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong